CLINICAL TRIAL: NCT03450252
Title: Distal Ventricular Pacing and Intraventricular Gradient Reduction for Symptomatic Relief in Drug Refractory Hypertrophic Cardiomyopathy Patients With Mid-cavity Obstruction
Brief Title: Pacemaker Therapy for Drug-refractory Symptoms in Mid-cavity Hypertrophic Cardiomyopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: V11_27 10 20
Record Dates: First submitted 2018-01-17; First posted 2018-03-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-02

CONDITIONS: Cardiomyopathy, Hypertrophic
Keywords: HCM; Mid-cavity; Pacing
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Intervention Model Description: Taking part in this study will involve recording the information at a pre-implant visit, a visit for cardiac pacemaker implantation and follow-up visits four and eight months later.
  At the pre-implant visit, participants will undergo assessment of symptoms, physical performance and blood test for a protein, Brain natriuretic peptide (BNP).
  During the pacemaker implantation, the investigators will record the pressures within the heart using a catheter during both active pacing and back-up pacing settings.
  The day after the pacemaker implant participants will undergo double-blind randomisation into either the treatment or non-treatment arm (active or back-up pacing respectively). At four months, cross-over takes place with assessment as above, before device reprogramming into either the treatment or non-treatment arm depending on which was completed first.
  At the end of the second four month period, participants will undergo repeat assessment as above. That will conclude the study.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active pacing (Experimental): Active ventricular pacing. The pacemaker is set-up with a short atrio-ventricular delay to allow for appropriate pacing capture of the ventricle.
  Interventions: Device: Active pacing
- Back-up pacing (Sham Comparator): Back-up pacing. The pacemaker is set-up to sense and pace only in the right atrium (AAI) without any pacing capacity in the ventricle.
  Interventions: Device: Back-up pacing

INTERVENTIONS:
Device: Active pacing — Ventricular pacing via the invasive haemodynamic study-defined optimal pacing site in order to relieve pressure gradient across the mid-cavity obstruction in mid-cavity obstructive variant hypertrophic cardiomyopathy.
  Arms: Active pacing
Device: Back-up pacing — Back-up pacing. The pacemaker is set-up to sense and pace only in the right atrium (AAI) without any pacing capacity in the ventricle.
  Arms: Back-up pacing

SUMMARY:
The main aim of this study is to assess the acute effects of a pacemaker on reducing abnormally high intracavity pressures in the hearts of patients with mid-cavity obstructive hypertrophic cardiomyopathy (HCM). During a 12-month period of double-blinded follow-up, descriptive data will be collected on patients symptomatic and physical performance during dichotomous pacemaker settings for 6-months each (active and back-up). The statistical information collected will be used to design a much larger research trial of patient benefit.

DETAILED DESCRIPTION:
Hypertrophic cardiomyopathy (HCM) is the most common inherited heart disease, affecting 1 in 500 of the general population. It is characterised by abnormal thickening of the heart muscle. The various patterns of thickening of the muscle in the main pumping chamber, or left ventricle (LV), can result in obstruction to blood flow within the heart, raising the pressures in the heart and placing extra strain on the heart muscle.

The obstruction can cause patients to suffer from symptoms such as shortness of breath and chest pain, along with poor exercise tolerance, and dizzy spells. In very symptomatic patients with the commonest type of obstruction, invasive procedures performed either via an open-heart or keyhole operation can reduce the increased basal septal muscle mass at the point of obstruction. However, in around 1 in 10 HCM patients, the obstruction is deep within the LV where a ring of thick muscle blocks blood flow when it contracts. These patients provide a challenge for doctors, as this type of obstruction is much less suitable for open heart or keyhole operation.

An alternative is to use a cardiac pacemaker to alter the timing of the contraction in the ring of thick muscle such that different parts of the ring contract at different times and thereby reduce obstruction to blood flow. The investigators' early experience with this new treatment shows that carefully placing the pacemaker wires can reduce the obstruction and improve patient symptoms.

Key questions of this research include:

* How much can optimal ventricular pacing reduce the obstruction by?
* How important is choosing which part of the heart the pacemaker activates first?
* Does reducing obstruction in this way make patients better in the short and long term?

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, >18 years.
2. Referred for PPM +/- ICD implantation for either primary prevention of sudden cardiac death or other indications such as heart block or obstructive physiology.
3. HCM patients with evidence of mid-cavity gradient demonstrated by echocardiography and gradient ≥30 mmHg confirmed by cardiac catheterisation at rest or with isoprenaline provocation.
4. All patients should be taking maximum tolerated doses of beta blockers or verapamil with or without disopyramide.
5. Symptoms refractory to optimum medical therapy as above, for example breathlessness, chest pain, dizziness, or syncope.

Exclusion Criteria:

1. Patients with multi-level obstruction, i.e. across the mid-cavity and outflow tract.
2. Patients with moderate or severe valvular stenosis or regurgitation.
3. Patients with a history of myocardial infarction or acute coronary syndrome.
4. Patients unable to provide informed consent.
5. Patients in atrial fibrillation.
6. Pregnancy.
7. Renal failure.
8. If considered unsuitable by clinician.
9. Patients already participating in trials involving invasive procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Invasive gradient (mmHg) | Measured during pacemaker implant. Pressure gradients will be measured at different pacing sites during the implant.
  Acute invasively defined gradient change in mmHg across the mid-cavity with optimal ventricular pacing setting

SECONDARY OUTCOMES:
Symptomatic assessment via SF36 questionnaire | Pre-implant, 4 months, and 8 months
  Generalised health related questionnaire
Symptomatic assessment via Kansas City Cardiomyopathy questionnaire | Pre-implant, 4 months, and 8 months
  Cardiomyopathy health related questionnaire
Symptomatic assessment via calculation of New York Heart Association (NYHA) functional class | Pre-implant, 4 months, and 8 months
  Classification of extent of heart failure
Exercise performance assessed by 6 minute walk test (6MWT) | Pre-implant, 4 months, and 8 months
  Sub-maximal exercise test
Exercise performance assessed by Cardiopulmonary exercise testing (CPET) stress echocardiography. | Pre-implant, 4 months, and 8 months
  Maximal exercise test with simultaneous echocardiography
Levels of Brain Natriuretic Peptide | Pre-implant, 4 months, and 8 months
  Protein associated with heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Saidi A Mohiddin, BSc, MBChB, FRCP, MD, Principal Investigator — Barts Health NHS Trust and Queen Mary University of London
Locations (1):
- Barts Heart Centre, London, Thames, United Kingdom

REFERENCES:
- [Derived] Malcolmson JW, Hughes RK, Husselbury T, Khan K, Learoyd AE, Lees M, Wicks EC, Smith J, Simms AD, Moon JC, Lopes LR, O'Mahony C, Sekhri N, Elliott PM, Petersen SE, Dhinoja MB, Mohiddin SA. Distal Ventricular Pacing for Drug-Refractory Mid-Cavity Obstructive Hypertrophic Cardiomyopathy: A Randomized, Placebo-Controlled Trial of Personalized Pacing. Circ Arrhythm Electrophysiol. 2024 Jul;17(7):e012570. doi: 10.1161/CIRCEP.123.012570. Epub 2024 Jun 19. PMID 39012930